CLINICAL TRIAL: NCT02105636
Title: An Open Label, Randomized Phase 3 Clinical Trial of Nivolumab vs Therapy of Investigator's Choice in Recurrent or Metastatic Platinum-refractory Squamous Cell Carcinoma of the Head and Neck (SCCHN)
Brief Title: Trial of Nivolumab vs Therapy of Investigator's Choice in Recurrent or Metastatic Head and Neck Carcinoma (CheckMate 141)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-141; 2013-003622-86 (EudraCT Number)
Record Dates: First submitted 2014-04-03; First posted 2014-04-07 (Estimated); Results first posted 2017-01-11 (Estimated); Last update posted 2022-10-05 (Actual); Status verified 2022-08

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Nivolumab; Cetuximab; Methotrexate; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Nivolumab (Experimental): Nivolumab 3mg/kg intravenous (IV) Solution for Injection every 2 weeks until disease progression
  Interventions: Drug: Nivolumab
- Arm B: Cetuximab/Methotrexate/Docetaxel (Active Comparator): Cetuximab intravenous (IV) Solution for Injection 400 mg/m2 (first dose) then 250 mg/m2 weekly until disease progression
  OR
  Methotrexate intravenous (IV) Solution for Injection 40 or 60 mg/m2 weekly until disease progression
  OR
  Docetaxel intravenous (IV) Solution for Injection 30 or 40 mg/m2 weekly until disease progression
  Interventions: Drug: Cetuximab; Drug: Methotrexate; Drug: Docetaxel

INTERVENTIONS:
Drug: Nivolumab
  Other Names: BMS-936558
  Arms: Arm A: Nivolumab
Drug: Cetuximab
  Arms: Arm B: Cetuximab/Methotrexate/Docetaxel
Drug: Methotrexate
  Arms: Arm B: Cetuximab/Methotrexate/Docetaxel
Drug: Docetaxel
  Arms: Arm B: Cetuximab/Methotrexate/Docetaxel

SUMMARY:
The purpose of this study is to find out whether Nivolumab will significantly improve overall survival as compared to therapy of investigator's choice in patients with recurrent or metastatic head and neck carcinoma.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Men and women ≥ 18 years of age with an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
* Histologically confirmed recurrent or metastatic SCCHN (oral cavity, pharynx, larynx), stage III/IV and not amenable to local therapy with curative intent (surgery or radiation therapy with or without chemotherapy)
* Tumor progression or recurrence within 6 months of last dose of platinum therapy in the adjuvant (ie with radiation after surgery), primary (ie, with radiation), recurrent, or metastatic setting
* Measurable disease by Computed tomography (CT) or Magnetic resonance imaging (MRI) per Response Evaluation Criteria In Solid Tumors (RECIST 1.1) criteria

Exclusion Criteria:

* Active brain metastases or leptomeningeal metastases are not allowed
* Histologically confirmed recurrent or metastatic carcinoma of the nasopharynx, squamous cell carcinoma of unknown primary, and salivary gland or non-squamous histologies (eg: mucosal melanoma) are not allowed
* Subjects with active, known or suspected autoimmune disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 361 (Actual)
Dates: Start 2014-05-29 (Actual); Primary Completion 2015-11-06 (Actual); Study Completion 2021-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (64):
- United States (15):
  - Stanford University Medical Center, Stanford, California
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Local Institution - 0001, Atlanta, Georgia
  - Local Institution - 0002, Chicago, Illinois
  - Local Institution - 0004, Metairie, Louisiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University Of Michigan, Ann Arbor, Michigan
  - Dumc, Durham, North Carolina
  - Local Institution - 0012, Columbus, Ohio
  - Local Institution - 0007, Pittsburgh, Pennsylvania
  - Vanderbilt Cancer Clinic, Nashville, Tennessee
  - Univ Of Tx. Md Anderson, Hoston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Local Institution - 0031, Milwaukee, Wisconsin
- Argentina (3):
  - Local Institution - 0015, Berazategui, Buenos Aires
  - Local Institution - 0013, San Miguel de Tucumán, Tucumán Province
  - Local Institution - 0014, Córdoba
- Brazil (3):
  - Local Institution - 0054, Ijuí, Rio Grande do Sul
  - Local Institution, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0055, São Paulo
- Canada (2):
  - Local Institution - 0038, Vancouver, British Columbia
  - Local Institution - 0045, London, Ontario
- France (3):
  - Local Institution, Lyon
  - Local Institution, Nice
  - Local Institution, Villejuif
- Germany (6):
  - Local Institution - 0047, Berlin
  - Local Institution - 0049, Bonn
  - Local Institution - 0048, Essen
  - Local Institution - 0052, Hamburg
  - Local Institution - 0046, Hanover
  - Local Institution - 0050, Würzburg
- Local Institution, Hong Kong, Hong Kong
- Italy (6):
  - Ist.Scient. Romagnolo Per Lo Studio E Cura Tumori, Meldola, FC
  - Local Institution, Milan, MI
  - Local Institution, Torino, TO
  - Local Institution, Milan
  - Local Institution, Napoli
  - Local Institution, Padua
- Japan (8):
  - Local Institution - 0056, Nagoya, Aichi-ken
  - Local Institution - 0060, Kashiwa, Chiba
  - Local Institution - 0062, Sapporo, Hokkaido
  - Local Institution - 0058, Kobe, Hyōgo
  - Local Institution - 0063, Takatsuki, Osaka
  - Local Institution - 0059, Sunto-gun, Shizuoka
  - Local Institution - 0057, Akashi, Hyogo
  - Local Institution - 0061, Tokyo
- Netherlands (3):
  - Local Institution, Amsterdam
  - Local Institution, Groningen
  - Local Institution, Leiden
- South Korea (2):
  - Local Institution - 0067, Seoul
  - Local Institution - 0066, Seoul
- Spain (4):
  - Local Institution - 0032, Barcelona
  - Local Institution - 0035, Barcelona
  - Local Institution - 0034, Madrid
  - Local Institution - 0033, Valencia
- Local Institution - 0051, Zurich, Switzerland
- Taiwan (2):
  - Local Institution - 0065, Tainan
  - Local Institution - 0064, Taipei
- United Kingdom (5):
  - Local Institution, London, Greater London
  - Local Institution, Manchester, Greater Manchester
  - Local Institution, Southampton, Hampshire
  - Local Institution, Metropolitan Borough of Wirral, Merseyside
  - Local Institution, Surrey, Surrey

REFERENCES:
- [Derived] Yen CJ, Kiyota N, Hanai N, Takahashi S, Yokota T, Iwae S, Shimizu Y, Hong RL, Goto M, Kang JH, Li WSK, Ferris RL, Gillison M, Endo T, Jayaprakash V, Tahara M. Two-year follow-up of a randomized phase III clinical trial of nivolumab vs. the investigator's choice of therapy in the Asian population for recurrent or metastatic squamous cell carcinoma of the head and neck (CheckMate 141). Head Neck. 2020 Oct;42(10):2852-2862. doi: 10.1002/hed.26331. Epub 2020 Jun 24. PMID 32583557
- [Derived] Saba NF, Blumenschein G Jr, Guigay J, Licitra L, Fayette J, Harrington KJ, Kiyota N, Gillison ML, Ferris RL, Jayaprakash V, Li L, Brossart P. Nivolumab versus investigator's choice in patients with recurrent or metastatic squamous cell carcinoma of the head and neck: Efficacy and safety in CheckMate 141 by age. Oral Oncol. 2019 Sep;96:7-14. doi: 10.1016/j.oraloncology.2019.06.017. Epub 2019 Jul 3. PMID 31422216
- [Derived] Cocks K, Contente M, Simpson S, DeRosa M, Taylor FC, Shaw JW. A Q-TWiST Analysis Comparing Nivolumab and Therapy of Investigator's Choice in Patients with Recurrent/Metastatic Platinum-Refractory Squamous Cell Carcinoma of the Head and Neck. Pharmacoeconomics. 2019 Aug;37(8):1041-1047. doi: 10.1007/s40273-019-00798-1. PMID 30972702
- [Derived] Pai SI, Faivre S, Licitra L, Machiels JP, Vermorken JB, Bruzzi P, Gruenwald V, Giglio RE, Leemans CR, Seiwert TY, Soulieres D. Comparative analysis of the phase III clinical trials of anti-PD1 monotherapy in head and neck squamous cell carcinoma patients (CheckMate 141 and KEYNOTE 040). J Immunother Cancer. 2019 Apr 3;7(1):96. doi: 10.1186/s40425-019-0578-0. PMID 30944020
- [Derived] Ferris RL, Blumenschein G Jr, Fayette J, Guigay J, Colevas AD, Licitra L, Harrington KJ, Kasper S, Vokes EE, Even C, Worden F, Saba NF, Docampo LCI, Haddad R, Rordorf T, Kiyota N, Tahara M, Lynch M, Jayaprakash V, Li L, Gillison ML. Nivolumab vs investigator's choice in recurrent or metastatic squamous cell carcinoma of the head and neck: 2-year long-term survival update of CheckMate 141 with analyses by tumor PD-L1 expression. Oral Oncol. 2018 Jun;81:45-51. doi: 10.1016/j.oraloncology.2018.04.008. Epub 2018 Apr 17. PMID 29884413
- [Derived] Kiyota N, Hasegawa Y, Takahashi S, Yokota T, Yen CJ, Iwae S, Shimizu Y, Hong RL, Goto M, Kang JH, Sum Kenneth Li W, Ferris RL, Gillison M, Namba Y, Monga M, Lynch M, Tahara M. A randomized, open-label, Phase III clinical trial of nivolumab vs. therapy of investigator's choice in recurrent squamous cell carcinoma of the head and neck: A subanalysis of Asian patients versus the global population in checkmate 141. Oral Oncol. 2017 Oct;73:138-146. doi: 10.1016/j.oraloncology.2017.07.023. Epub 2017 Sep 1. PMID 28939066
- [Derived] Harrington KJ, Ferris RL, Blumenschein G Jr, Colevas AD, Fayette J, Licitra L, Kasper S, Even C, Vokes EE, Worden F, Saba NF, Kiyota N, Haddad R, Tahara M, Grunwald V, Shaw JW, Monga M, Lynch M, Taylor F, DeRosa M, Morrissey L, Cocks K, Gillison ML, Guigay J. Nivolumab versus standard, single-agent therapy of investigator's choice in recurrent or metastatic squamous cell carcinoma of the head and neck (CheckMate 141): health-related quality-of-life results from a randomised, phase 3 trial. Lancet Oncol. 2017 Aug;18(8):1104-1115. doi: 10.1016/S1470-2045(17)30421-7. Epub 2017 Jun 23. PMID 28651929
- [Derived] Ferris RL, Blumenschein G Jr, Fayette J, Guigay J, Colevas AD, Licitra L, Harrington K, Kasper S, Vokes EE, Even C, Worden F, Saba NF, Iglesias Docampo LC, Haddad R, Rordorf T, Kiyota N, Tahara M, Monga M, Lynch M, Geese WJ, Kopit J, Shaw JW, Gillison ML. Nivolumab for Recurrent Squamous-Cell Carcinoma of the Head and Neck. N Engl J Med. 2016 Nov 10;375(19):1856-1867. doi: 10.1056/NEJMoa1602252. Epub 2016 Oct 8. PMID 27718784
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Nivolumab 3mg/kg: Nivolumab was provided at a dose of 3 milligrams/kilogram (mg/kg) using an intravenous (IV) solution for Injection every 2 weeks until disease progression.
- Investigators Choice: Participants were provided a dose of Cetuximab intravenous (IV) solution for injection at a dose of 400 milligrams per square meter (mg/m^2) for the first dose followed that a doses of 250 mg/m^2 weekly until disease progression OR a Methotrexate intravenous (IV) solution for Injection at a dose of 40 or 60 mg/m^2 weekly until disease progression OR a Docetaxel intravenous (IV) solution for Injection at a dose of 30 or 40 mg/m^2 weekly until disease progression. The decision regarding which treatment the participant received was at the discretion of the investigator and referred to as Investigators Choice
Period: Pre-Treatment
Arm/Group | Nivolumab 3mg/kg | Investigators Choice
Started (Started = Randomized) | 240 | 121
Completed (Completed = Entering treatment) | 236 | 111
Not Completed | 4 | 10
Not completed — Disease Progression | 1 | 0
Not completed — Participant request to discontinue study treatment | 1 | 2
Not completed — Participant withdrew consent | 0 | 6
Not completed — Participant no longer meets study criteria | 2 | 2
Period: Treatment
Arm/Group | Nivolumab 3mg/kg | Investigators Choice
Started | 236 | 111
Completed | 1 | 0
Not Completed | 235 | 111
Not completed — Study Drug Toxicity | 14 | 10
Not completed — Adverse event unrelated to study drug | 19 | 3
Not completed — Participant request to discontinue study treatment | 8 | 6
Not completed — Participant withdrew consent | 5 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Maximum Clinical Benefit | 1 | 3
Not completed — Poor/Non-compliance | 0 | 1
Not completed — Participant no longer meets study criteria | 1 | 0
Not completed — Other reasons | 1 | 0
Not completed — Disease Progression | 185 | 87

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nivolumab 3mg/kg | Investigators Choice | Total
Number analyzed (Participants) | 240 | 121 | 361
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.0 (10.15) | 59.4 (11.00) | 59.1 (10.43)
Age, Customized [Number; unit: Participants]
  < 65 years | 172 | 76 | 248
  >=65 and <75 years | 56 | 39 | 95
  >=75 years | 12 | 6 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 18 | 61
  Male | 197 | 103 | 300
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 196 | 104 | 300
  Black or African American | 10 | 3 | 13
  Asian | 29 | 14 | 43
  Other | 5 | 0 | 5
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic/Latino | 9 | 4 | 13
  Not Hispanic/Latino | 132 | 60 | 192
  Not Reported | 99 | 57 | 156

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to the date of death from any cause. Participants were censored at the date they were last known to be alive and at the date of randomization if they were randomized but had no follow-up. Median OS time was calculated using Kaplan-Meier (KM) method.
Time Frame: From date of randomization to date of death (Up to approximately 18 months)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab 3mg/kg | Investigators Choice
Number analyzed (Participants) | 240 | 121
Months | 7.49 [5.49 to 9.10] | 5.06 [4.04 to 6.05]
Statistical Analysis 1: Comparison: Nivolumab 3mg/kg vs Investigators Choice; Stratified Cox proportional hazard model. HR = Nivolumab over investigator's choice therapy (Cetuximab, Methotrexate, or Docetaxel); Test type: Superiority; p = 0.0101, Log Rank — Log-rank Test stratified by prior treatment with cetuximab (yes, no) as entered into the Interactive Voice Response System (IVRS). For OS the boundary for statistical significance requires the p-value to be less than 0.0227; Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.53 to 0.92] — Hazard ratio (HR) and the corresponding Confidence Interval (CI) were estimated in a stratified Cox proportional hazards model for distribution of OS in each randomized arm

2. Secondary Outcome: Investigator-Assessed Progression-Free Survival (PFS)
Description: PFS was defined as the time between the date of randomization and the first date of documented progression, as determined by the investigator (as per Response Evaluation Criteria In Solid Tumors (RECIST1.1)), or death due to any cause, whichever occurs first. Progressive Disease: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. The sum must demonstrate an absolute increase of at least 5mm. Participants who:
  * Die without a reported progression were considered to have progressed on the date of their death.
  * Did not progress or die were censored on the date of their last evaluable tumor assessment.
  * Without any on study tumor assessments and did not die were censored on their date of randomization.
  * Received subsequent systemic anti-cancer therapy prior to documented progression were censored at the date of the last tumor assessment prior to the initiation of the new therapy.
Time Frame: From date of randomization to date of disease progression or death, whichever occurs first (Up to approximately 87 months)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab 3mg/kg | Investigators Choice
Number analyzed (Participants) | 240 | 121
Months | 2.04 [1.91 to 2.14] | 2.33 [1.94 to 3.06]
Statistical Analysis 1: Comparison: Nivolumab 3mg/kg vs Investigators Choice; Test type: Superiority; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.68 to 1.10] — Number of responders (CR +PR) over number of participants

3. Secondary Outcome: Investigator-Assessed Objective Response Rate (ORR)
Description: ORR was defined as the percentage of randomized participants who achieved a best response of complete response (CR) or partial response (PR) using the RECIST1.1 criteria as per investigator assessment. Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions.
Time Frame: From date of randomization to date of disease progression or study drug is discontinued, whichever occurs first (Up to approximately 87 months)
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Nivolumab 3mg/kg | Investigators Choice
Number analyzed (Participants) | 240 | 121
Percentage of Participants | 13.3 [9.3 to 18.3] | 5.8 [2.4 to 11.6]
Statistical Analysis 1: Comparison: Nivolumab 3mg/kg vs Investigators Choice; Test type: Superiority; Difference in ORR = 7.6, 95% CI 2-sided [1.5 to 13.6] — Stratum adjusted difference in response rates (Nivolumab - Investigators Choice) based on the Cochran-Mantel-Haenszel method of weighting
Statistical Analysis 2: Comparison: Nivolumab 3mg/kg vs Investigators Choice; Test type: Superiority; CMH Estimate of Common Odds Ratio = 2.49, 95% CI 2-sided [1.07 to 5.82] — Stratified by Prior Cetuximab (yes, no) as recorded in the IVRS. Stratum adjusted odds ratio (Nivolumab - Investigators Choice) using Mantel-Haenszel Method

4. Post Hoc Outcome: Overall Survival (OS) - Extended Collection
Description: OS was defined as the time from randomization to the date of death from any cause. Participants were censored at the date they were last known to be alive and at the date of randomization if they were randomized but had no follow-up. Median OS time was calculated using Kaplan-Meier (KM) method.
  Note: This outcome measure represents an updated version of the primary endpoint to include additional data collection that has occurred after the primary completion date. (Assessments were made until 10-Sep-2021)
Time Frame: From date of randomization to date of death (Up to approximately 87 months)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab 3mg/kg | Investigators Choice
Number analyzed (Participants) | 240 | 121
Months | 7.72 [5.68 to 8.74] | 5.06 [4.04 to 6.24]
Statistical Analysis 1: Comparison: Nivolumab 3mg/kg vs Investigators Choice; Test type: Superiority; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.54 to 0.85] — Stratified Cox proportional hazards model. Hazard ratio of nivolumab to investigator's choice therapy

ADVERSE EVENTS:
Time Frame: Adverse Events and Serious Adverse Events were monitored from first dose to 100 days post last dose (Up to a maximum of approximately 70 months). Participants were assessed for All Cause Mortality from their date of randomization until the study was completed (up to approximately 87 months)
Description: The number at Risk for All-Cause Mortality represents all Randomized Participants. The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication
Groups:
- Investigator Choice: Participants were provided a dose of Cetuximab intravenous (IV) solution for injection at a dose of 400 milligrams per square meter (mg/m^2) for the first dose followed that a doses of 250 mg/m^2 weekly until disease progression OR a Methotrexate intravenous (IV) solution for Injection at a dose of 40 or 60 mg/m^2 weekly until disease progression OR a Docetaxel intravenous (IV) solution for Injection at a dose of 30 or 40 mg/m^2 weekly until disease progression. The decision regarding which treatment the participant received was at the discretion of the investigator and referred to as Investigators Choice
Arm/Group | Nivolumab 3mg/kg | Investigator Choice
All-Cause Mortality (participants affected / at risk) | 220/240 | 119/121
Serious Adverse Events (participants affected / at risk) | 165/236 | 87/111
Other Adverse Events (participants affected / at risk) | 210/236 | 108/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab 3mg/kg (N=236) | Investigator Choice (N=111)
Anaemia (Blood and lymphatic system disorders) | 2 | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Atrial flutter (Cardiac disorders) | 1 | 1
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 3
Cardiac failure (Cardiac disorders) | 2 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Cardiovascular disorder (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Hypophysitis (Endocrine disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Secondary adrenocortical insufficiency (Endocrine disorders) | 1 | 0
Secondary hypothyroidism (Endocrine disorders) | 1 | 0
Blindness unilateral (Eye disorders) | 1 | 0
Visual acuity reduced (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 3
Ascites (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 3
Dysphagia (Gastrointestinal disorders) | 3 | 3
Gastric disorder (Gastrointestinal disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Oesophageal stenosis (Gastrointestinal disorders) | 1 | 0
Parotid gland haemorrhage (Gastrointestinal disorders) | 1 | 0
Pneumoperitoneum (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 1
Tongue haemorrhage (Gastrointestinal disorders) | 2 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 2
Catheter site pain (General disorders) | 1 | 0
Chills (General disorders) | 1 | 1
Death (General disorders) | 1 | 0
Face oedema (General disorders) | 1 | 1
Fatigue (General disorders) | 3 | 1
General physical health deterioration (General disorders) | 1 | 0
Localised oedema (General disorders) | 1 | 0
Malaise (General disorders) | 0 | 2
Mucosal inflammation (General disorders) | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 1
Pyrexia (General disorders) | 5 | 4
Ulcer haemorrhage (General disorders) | 1 | 0
Bile duct stenosis (Hepatobiliary disorders) | 1 | 0
Contrast media allergy (Immune system disorders) | 0 | 1
Eosinophilic granulomatosis with polyangiitis (Immune system disorders) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 1
Device related infection (Infections and infestations) | 1 | 1
Gastrointestinal infection (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 2 | 0
Localised infection (Infections and infestations) | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 3 | 3
Lymphangitis (Infections and infestations) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 1 | 1
Osteomyelitis (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 17 | 5
Pneumonia bacterial (Infections and infestations) | 1 | 0
Pneumonia pseudomonal (Infections and infestations) | 0 | 1
Purulent discharge (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 5 | 1
Sepsis (Infections and infestations) | 6 | 4
Septic shock (Infections and infestations) | 3 | 1
Sinusitis (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 0 | 1
Systemic infection (Infections and infestations) | 1 | 0
Tracheitis (Infections and infestations) | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 4 | 0
Vascular device infection (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 3 | 2
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 3 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 | 1
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Shunt thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Tracheostomy malfunction (Injury, poisoning and procedural complications) | 1 | 0
Vascular pseudoaneurysm ruptured (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1
Wound haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
General physical condition abnormal (Investigations) | 0 | 1
Liver function test abnormal (Investigations) | 1 | 0
Liver function test increased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 0 | 1
Transaminases increased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 4 | 1
Dehydration (Metabolism and nutrition disorders) | 4 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 1 | 1
Hyperamylasaemia (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 3 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 1
Hypophagia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Head and neck cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 94 | 55
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 1
Dizziness (Nervous system disorders) | 0 | 2
Encephalopathy (Nervous system disorders) | 1 | 0
Focal dyscognitive seizures (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Hydrocephalus (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 1
Radiculopathy (Nervous system disorders) | 0 | 1
Speech disorder (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 1
Device leakage (Product Issues) | 1 | 0
Device occlusion (Product Issues) | 0 | 1
Agoraphobia (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 | 2
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 10 | 4
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Stridor (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatomyositis (Skin and subcutaneous tissue disorders) | 0 | 1
Skin mass (Skin and subcutaneous tissue disorders) | 1 | 0
Skin toxicity (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 0 | 1
Haemorrhage (Vascular disorders) | 2 | 0
Hypertensive urgency (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Hypovolaemic shock (Vascular disorders) | 0 | 1
Shock haemorrhagic (Vascular disorders) | 1 | 0
Superior vena cava syndrome (Vascular disorders) | 1 | 0
Venous thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab 3mg/kg (N=236) | Investigator Choice (N=111)
Anaemia (Blood and lymphatic system disorders) | 53 | 42
Neutropenia (Blood and lymphatic system disorders) | 2 | 9
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 6
Tachycardia (Cardiac disorders) | 7 | 7
Hypothyroidism (Endocrine disorders) | 21 | 7
Lacrimation increased (Eye disorders) | 1 | 6
Constipation (Gastrointestinal disorders) | 43 | 21
Diarrhoea (Gastrointestinal disorders) | 47 | 27
Dry mouth (Gastrointestinal disorders) | 8 | 8
Dyspepsia (Gastrointestinal disorders) | 7 | 6
Dysphagia (Gastrointestinal disorders) | 30 | 17
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 8
Nausea (Gastrointestinal disorders) | 55 | 37
Stomatitis (Gastrointestinal disorders) | 14 | 12
Vomiting (Gastrointestinal disorders) | 28 | 16
Asthenia (General disorders) | 27 | 24
Face oedema (General disorders) | 11 | 8
Fatigue (General disorders) | 67 | 37
Mucosal inflammation (General disorders) | 11 | 19
Oedema peripheral (General disorders) | 19 | 5
Pyrexia (General disorders) | 37 | 16
Oral candidiasis (Infections and infestations) | 11 | 6
Pneumonia (Infections and infestations) | 16 | 5
Respiratory tract infection (Infections and infestations) | 6 | 6
Alanine aminotransferase increased (Investigations) | 9 | 6
Aspartate aminotransferase increased (Investigations) | 14 | 6
Blood alkaline phosphatase increased (Investigations) | 18 | 3
Lipase increased (Investigations) | 13 | 2
Lymphocyte count decreased (Investigations) | 8 | 6
Weight decreased (Investigations) | 35 | 19
White blood cell count decreased (Investigations) | 3 | 8
Decreased appetite (Metabolism and nutrition disorders) | 46 | 21
Hypercalcaemia (Metabolism and nutrition disorders) | 17 | 8
Hyperglycaemia (Metabolism and nutrition disorders) | 16 | 9
Hypoalbuminaemia (Metabolism and nutrition disorders) | 12 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 11 | 7
Hyponatraemia (Metabolism and nutrition disorders) | 25 | 15
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 17 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 17 | 9
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 | 8
Dizziness (Nervous system disorders) | 9 | 7
Headache (Nervous system disorders) | 23 | 4
Neuropathy peripheral (Nervous system disorders) | 6 | 9
Paraesthesia (Nervous system disorders) | 4 | 6
Anxiety (Psychiatric disorders) | 9 | 9
Depression (Psychiatric disorders) | 12 | 3
Insomnia (Psychiatric disorders) | 13 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 37 | 13
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 32 | 12
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 11
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 | 6
Productive cough (Respiratory, thoracic and mediastinal disorders) | 14 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 16
Dry skin (Skin and subcutaneous tissue disorders) | 14 | 12
Erythema (Skin and subcutaneous tissue disorders) | 3 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 23 | 1
Rash (Skin and subcutaneous tissue disorders) | 22 | 6
Hypertension (Vascular disorders) | 16 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.